CLINICAL TRIAL: NCT00639197
Title: UGIST Pilot Trial: Ultrasound Guided Internal Jugular Short-Term Central Venous Catheters Tunneling. Does it Reduce the Technical Difficulty and Mechanical Complications?
Brief Title: UGIST: Ultrasound Guided Internal Jugular Short-Term Central Venous Catheters Tunneling
Acronym: UGIST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: SALAH ALI TAQI, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08-007
Record Dates: First submitted 2008-03-11; First posted 2008-03-20 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-03

CONDITIONS: Infection; Bacteremia
Keywords: Tunneling; Short term; central venous catheters; Ultrasound Guided; Internal jugular; Assess safety and improve technical difficulty
MeSH Terms: conditions — Infections; Bacteremia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): To Tunnel
  Interventions: Procedure: To tunnel
- 2 (Active Comparator): Not to tunnel
  Interventions: Procedure: Standard (not to tunnel)

INTERVENTIONS:
Procedure: To tunnel — Using the standard Seldinger technique and under the guidance of ultrasound, the catheter will pass through a 3-5cm subcutaneous tunnel before it is eventually secured to reside at the internal jugular vein.
  Arms: 1
Procedure: Standard (not to tunnel) — Using the standard Seldinger technique and under the guidance of ultrasound, the catheter is secured to reside at the internal jugular vein, without a subcutaneous tunnel.
  Arms: 2

SUMMARY:
The purpose of the study is to determine if tunneling standard short-term central lines for a short distance under the skin, with the assistance of ultrasound imaging, reduces the risk of central line infections for catheters placed in the neck vein.

Previous work has shown that these lines can be tunneled without ultrasound guidance. We wish to determine if the use of ultrasound makes the tunneling procedure safer and easier.

DETAILED DESCRIPTION:
More than 250,000 vascular catheter-related bloodstream infections occur annually in the USA with a mortality ranging from 12% to 25% in critically ill patients.

It is also widely accepted that the internal jugular site is associated with a higher risk of catheter related infection if compared with the subclavian site.

Therefore, the benefit of catheter tunneling was best seen at the internal jugular site as described by J F Timsit in 1996 in his prospective randomized multicentre study where it significantly decreased the rate of catheter related sepsis from 11.4% to 3.4%.

At the same time, tunneling catheters did not increase the rate of mechanical complications such as pneumothorax, hematoma, or arterial puncture, but it almost doubled the rate of technical difficulties, such as problems with advancing the catheter or multiple puncture sites, at that time it was a blind technique.

Now, and with the introduction of the ultrasound guidance in our routine central line insertions, we would like to evaluate its benefit in reducing the technical difficulty and mechanical complications that used to be encountered while tunneling the short term central venous catheters at the internal jugular site.

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients.
* Likely to need the line for 48 hours.
* Standard central venous catheter.

Exclusion Criteria:

* Mechanical impedance (e.g C-spine protection).
* Absent Internal jugular vessel on U/S.
* Previous line still in place.
* Presence of overlying skin or tissue infection or mass.
* Tricuspid valve vegetation.
* Tumor extending to the right atrium.
* Persistent coagulopathy.
* Newly inserted Pacemaker leads.
* Recent carotid endarterectomy on same side.
* No ultrasound facility available.
* Patients requiring special lines (e.g. Dialysis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-03; Primary Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Reduction in Technical difficulty | 6-8 weeks for the whole 20 pts.

SECONDARY OUTCOMES:
Signs of line related blood stream infection/bacteremia. | 6-8 weeks for all 20 pts.

CONTACTS AND LOCATIONS:
Overall Officials: Salah A Taqi, MBChB, Principal Investigator — McMaster Health Sciences
Locations (1):
- Hamilton Health Sciences Corporation, Hamilton, Ontario, Canada